CLINICAL TRIAL: NCT04826315
Title: A Patient-Caregiver Behavioral Intervention for Older Adults With Cancer and Mild Cognitive Impairment
Brief Title: Cancer and Mild Cognitive Impairment a Patient-Caregiver Behavioral Intervention
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study halted prematurely, prior to enrollment of first participant
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00107680
Record Dates: First submitted 2021-03-29; First posted 2021-04-01 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Cancer; Cognitive Impairment
Keywords: Aging; Behavioral Intervention; Mental Health; Communication
MeSH Terms: conditions — Neoplasms; Cognitive Dysfunction; Psychological Well-Being; Communication | interventions — Coatomer Protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient Caregiver Dyad (Experimental): Participants who are 65 years or older with cancer and mild cognitive impairment with their caregiver.
  Interventions: Behavioral: COPE +

INTERVENTIONS:
Behavioral: COPE + — Six sixty minute sessions that teaches participants distress and communication coping skills.

SUMMARY:
The purpose of this study is to see whether programs that include both a patient and their spouse or a patient and family caregiver (known as a dyad) are helpful for families in which one member of the dyad has cancer and mild memory difficulties and/or concerns. Participant and their spouse or participant and their family caregiver will have six, 60-minute video-conference sessions which will be scheduled at their convenience. The investigator will loan participants a tablet computer (iPad) to use for videoconferencing and train the participant in its use. Participant and their spouse or participant and their family caregiver will complete three assessments - one before starting the sessions, one after the sixth session, and one after 1 month. Each assessment will include surveys, which the participant will complete separately from their spouse or family caregiver. For most people, it will take upwards of 2 - 4 months to complete this study.

ELIGIBILITY:
Inclusion Criteria:

Patient inclusion criteria include:

1. Patients with Stage I-IV breast, colon, rectal, or lung cancer (newly diagnosed within 6 months; age 65 or older.
2. Participants must be living at home (either in her/his own home).
3. Participants must be fluent in English and able to learn basic skills for using a tablet computer to conduct videoconference treatment sessions.
4. Exhibit Mild Cognitive Impairment.
5. Have an informal family caregiver.

Inclusion Criteria:

(Partner or family member) inclusion criteria include:

1. Caregivers are 18 older.
2. Be fluent in English and able to learn basic skills for using a tablet computer to conduct videoconference treatment sessions.
3. Either co-reside with the patient or spend at least 3-4 hours day caregiving.
4. Not exhibit cognitive impairment.

Exclusion Criteria for both patients and caregivers:

1. Participant has visual or hearing impairments that preclude participation.
2. Participant has dementia and do not have the capacity to participate.
3. Have a serious untreated psychiatric illness as documented in medical chart review.
4. The patient and the caregiver score less than a 3 on the National Comprehensive Cancer Network (NCCN) Distress Thermometer (DT) on a scale 0 to 10 to screen for distress.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-15 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Number of completed sessions as measured by enrollment log | Up to 10 weeks
Number of participants who are satisfied with the intervention as measured by a score of 24 or greater on the CSQ-8 | Up to 10 weeks.
  The Client Satisfaction Questionnaire (CSQ-8) is a self report measure of satisfaction with health and behavioral services received. The CSQ-8 is measured on a four point Likert scale from 1 "Quite Dissatisfied" to 4 "Very Satisfied." Scores range from 8-32, with higher values indicating higher satisfaction.

SECONDARY OUTCOMES:
Change in Distress as measured by the DASS-21 | Up to 10 weeks.
  The Depression, Anxiety, and Stress Scale (DASS-21) measure will be used for rating general distress across three emotional states of depression, anxiety, and stress. The measure has a total of 21 items. Scores range from 0- 63, with higher scores indicating greater distress.
Change in Quality of Life as measured by the FACT-G | Up to 10 weeks.
  The Functional Assessment of Cancer Therapy: General (FACT-G) measure will be used for rating quality of life. The measure has a total of 27 items. Scores range from 0-108, with higher scores indicating greater quality of life.
Change in Communication Patterns as measured by the CPQ-SF | Up to 10 weeks.
  The Communication Patterns Questionnaire Short-Form (CPQ-SF) will be used for rating communication patterns in a relationship. The measure has a total of 11 items. Scores range from 11-99, higher scores indicate a greater likelihood of using a particular communication pattern during conflict interactions.
Change in Relationship Satisfaction as measured by the Mutuality Scale of the Family Care Inventory | Up to 10 weeks.
  The Mutuality Scale of the Family Care Inventory will be used for rating mutual concerns and overall relationship satisfaction. The measure consists of 15 items. Scores range from 0-60, higher scores indicate greater relationship satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine Ramos, Ph.D., Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No